CLINICAL TRIAL: NCT05229315
Title: PD-1 Immune Checkpoint Inhibitor Combined With Intensity Modulated Radiation Therapy in the Treatment of Intermediate-risk Nasopharyngeal Carcinoma (T2-3N0 or T1-2N1 and EBV-DNA≤4000 Copy/ml),A Single-arm, Phase II Clinical Trial
Brief Title: PD-1 Combined With Intensity Modulated Radiation Therapy in the Treatment of Intermediate-risk Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: XIANG YANQUN (Other)
Responsible Party: Sponsor-Investigator, XIANG YANQUN, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-292-01
Record Dates: First submitted 2022-01-25; First posted 2022-02-08 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Nasopharyngeal Carcinoma; T2-3N0 or T1-2N1; EBV-DNA≤4000 Copy/ml
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 Immune Checkpoint Inhibitor Combined With Intensity Modulated Radiation Therapy (Experimental): Intensity modulated radiation therapy combined with toripalimab in the treatment of nasopharyngeal carcinoma，once every 2 weeks, 10 cycles in total
  Interventions: Drug: Toripalimab; Procedure: Intensity modulated radiotherapy

INTERVENTIONS:
Drug: Toripalimab — PD-1 Immune Checkpoint Inhibitor Combined With IMRT,used at 2 weeks before radiotherapy, once every 2 weeks, 10 cycles in total
  Other Names: Programmed cell death protein 1(PD-1)；Immune checkpoint inhibitors（ICIs)
Procedure: Intensity modulated radiotherapy — Intensity modulated radiotherapy

SUMMARY:
To evaluate the safety and efficacy of PD-1 immune checkpoint inhibitor combined with intensity modulated radiation therapy in the treatment of intermediate-risk nasopharyngeal carcinoma (T2-3N0 or T1-2N1 stage and EBV-DNA≤4000 copy/ml).

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of PD-1 immune checkpoint inhibitor combined with intensity modulated radiation therapy in the treatment of intermediate-risk nasopharyngeal carcinoma (T2-3N0 or T1-2N1 stage and EBV-DNA≤4000 copy/ml).The primary end point is safety, the secondary end points are short-term efficacy,overall survival (OS), progression-free survival (PFS),Distant metastasis-free survival(DMFS),adverse effects ,quality of life and immune status assessment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients who have not received radiotherapy or chemotherapy
* Pathologically diagnosed as non-keratinizing nasopharyngeal carcinoma (differentiated or undifferentiated, WHO classification type II or type III).
* T2-3N0 or T1-2N1 stage and EBV-DNA≤4000 copy/ml (AJCC 8th version) and EBV-DNA≤4000copies/ml
* Male or non-pregnant female
* Age between 18 and 65
* Eastern Cooperative Oncology Group（ECOG）score of 0-1.
* Hemoglobin (HGB) ≥90 g/L, white blood cell (WBC) ≥4×109/L, platelet (PLT) ≥100×109/L.
* Liver function: Alanine aminotransferase (ALT), aspartate aminotransferase (AST) <2.0 times the upper limit of normal (ULN); total bilirubin <2.0×ULN.
* Renal function: creatinine clearance rate ≥60ml/min or serum creatinine <1.5×ULN.
* The patient has signed the informed consent

Exclusion Criteria:

* The pathology is keratinizing squamous cell carcinoma (WHO classification is type I).
* Patients with recurrence and distant metastasis.
* Patients who have undergone radiotherapy or chemotherapy.
* Active hepatitis B (HBV-DNA≥500).
* Patients with autoimmune diseases.
* Patients with HIV infection.
* At the same time suffering from other uncontrolled serious diseases.
* Persons with abnormal functions of the heart, brain, lungs and other important organs.
* Age> 65 years.
* pregnancy or breast feeding.
* Persons with personality or mental illness, without or with limited capacity for civil conduct

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-03-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Recent evaluation: 3 months after the end of treatment；Long-term follow-up: 1~5 years after the end of treatment
  The severity of adverse events will be determined by the investigator based on CTCAE v 5.0

SECONDARY OUTCOMES:
overall survival (OS) | 2 years
  Patients in clinical trials were randomized to the time of death from any cause
progression-free survival (PFS) | 2 years
  The time from the commencement of a randomized clinical trial to the progression of tumorigenesis (in any respect) or death from any cause
Distant metastasis-free survival(DMFS) | 2 years
  Patients in clinical trials were randomized to the time of distant metastasis
Response rate (based on RECIST ver1.1) | Recent evaluation: 3 months after the end of treatment；Long-term follow-up: 1~5 years after the end of treatment
  According to the remission assessment criteria of solid tumors，divided into CR, PR, SD, PD.
  CR(complete response) All target lesions disappeared and no new lesions appeared PR ( partial response) reduction of the sum of the largest diameters of target lesions by ≥30%) SD(stable disease)the sum of the largest diameters of target lesions does not shrink to PR, or increases to PD PD(progressive disease) The sum of the largest diameters of target lesions increases by at least 20%, or new lesions appear

CONTACTS AND LOCATIONS:
Overall Officials: Yanqun Xiang, Dr, Principal Investigator — Sun Yat-sen University
Locations (1):
- Yanqun Xiang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes